CLINICAL TRIAL: NCT06672926
Title: NEWPROMRI-PATHWAY - A New Prostate Magnetic Resonance Imaging (MRI) Pathway
Acronym: NEWPROMRI
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospitals of North Midlands NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 3320
Record Dates: First submitted 2024-10-25; First posted 2024-11-04 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer; MRI
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prostate cancer is the second most common cancer in men worldwide. The demand for magnetic resonance imaging (MRI) to diagnose and manage prostate cancer is continually growing. There is, however, a severe global shortage of radiologists who review and make decisions on prostate scans. This shortage causes compromises that are inefficient and negatively affect care provision, patient outcomes, and patient experiences. Two key examples of these compromises are that every patient receives a gadolinium contrast injection during a prostate MRI scan and patients often require multiple imaging appointments. If radiologists' knowledge of making prostate MRI decisions around these compromises could be harnessed and passed to radiographers (who are trained to acquire the MRIs but currently do not review them) with a computerised system to support clinical decision-making, this would have enormous potential to improve the diagnosing and managing prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* MRI radiographers in University Hospitals of North Midlands (UHNM) and or University Hospitals of Derby and Burton (UHDB) with over 5 years' experience in MRI of the prostate.
* Radiographers from UHNM or UHDB who have completed an online and hands on study specific training materials before the testing phase.
* Retrospective data of 800 patients each from UHNM and UHDB who have had mpMRI and went on to have a biopsy.

Exclusion Criteria:

* Non-MRI radiographers.
* Radiographers who did not completed an online and hands on study specific training materials before the testing phase.
* Non-mpMRI.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Uro-radiologists will be asked to take part, along with radiographers and members of a prostate cancer charity group
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Use of Gadolinium Based Contrast Agent (GBCA) injection | 12 months
  Equivalence between radiographers and radiologists in deciding when Gadolinium Based Contrast Agent (GBCA) injection is required in prostate MRI scans. This is by comparing radiographers' diagnoses (decisions on whether GBCA injection would have been required) with radiologists' decisions to determine equivalence in prostate cancer diagnosis using prostate MRI.
Application of WB-MRI | 12 months
  Equivalence between radiographers and radiologists in deciding when WB-MRI is required in prostate MRI scans. This is by comparing radiographers' decisions (decisions on whether WB-MRI would have been required) with radiologists' decisions to determine equivalence in prostate cancer diagnosis using prostate MRI.
Radiographers opinions | 12 months
  The Decisional Conflict Scale (DCS) will be used to capture radiographers' opinions on how they felt about the tasks and support they are given during their preparation and afterward

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of North Midlands NHS Trust, Stoke-on-Trent, Staffordshire, United Kingdom